CLINICAL TRIAL: NCT04031430
Title: PREMOM II: Pregnancy Remote Monitoring of Women with Gestational Hypertensive Disorders
Brief Title: PREMOM-II: Pregnancy Remote Monitoring of Women with Gestational Hypertensive Disorders
Acronym: PREMOM-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Universitaire Ziekenhuizen KU Leuven (Other); AZ Sint-Jan AV (Other); AZ Sint-Lucas Brugge (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Wilfried Gyselaers, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREMOM-II
Record Dates: First submitted 2018-11-21; First posted 2019-07-24 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Gestational Hypertension
Keywords: remote monitoring; gestational hypertensive disorders; pregnancy outcomes
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- telemonitoring group (TM) (Experimental): telemonitoring group (TM)
  Interventions: Device: Telemonitoring
- Patient self-monitoring group (PSM) (Active Comparator): Patient self-monitoring group (PSM)
  Interventions: Device: Telemonitoring
- control group (CC) (No Intervention): No intervention
- CAPROM - Group 1 (Experimental): pregnant women randomly assigned to the TM group of PREMOM II
  Interventions: Other: Longitudinal CV profiling during pregnancy and before and after the start/switch of antihypertensive medication
- CAPROM - Group 2 (Experimental): pregnant women followed-up via TM group as part of their usual care
  Interventions: Other: CV profiling before and after the start/switch of antihypertensive medication

INTERVENTIONS:
Device: Telemonitoring — Women who are allocated to the PSM groep, will receive a connected blood pressure monitor. They have to measure their blood pressure twice a day and fill in their weight once a week in the App. These data are automatically transmitted via Bluetooth and Wi-Fi to the hospital, but the caregiver will not see those data, and can not react to it.
  Arms: Patient self-monitoring group (PSM); telemonitoring group (TM)
Other: Longitudinal CV profiling during pregnancy and before and after the start/switch of antihypertensive medication — Longitudinal CV profiling during pregnancy and before and after the start/switch of antihypertensive medication Registration of medication usage in the Medisafe app Assessment of their beliefs about medicine in general and during pregnancy and their perceptions regarding medication adherence by means of the 'Beliefs about Medicine Questionnaire' and the 'Probabilistic Medication Adherence Scale' at baseline and postpartum.
  Arms: CAPROM - Group 1
Other: CV profiling before and after the start/switch of antihypertensive medication — CV profiling before and after the start/switch of antihypertensive medication Registration of medication usage in the Medisafe app Assessment of their beliefs about medicine in general and during pregnancy and their perceptions regarding medication adherence by means of the 'Beliefs about Medicine Questionnaire' and the 'Probabilistic Medication Adherence Scale' at baseline and postpartum.
  Arms: CAPROM - Group 2

SUMMARY:
The goal of this project is thoroughly evaluate the added value of telemonitoring (TM) program for women at risk for gestational hypertensive disorders (GHD), by investigating it impact on prenatal follow-up, health outcomes for mother and child, costs and satisfaction, and by specifically investigating what are the major contributors to this added value.

A substudy (CAPROM) will be conducted at the Department of Obstetrics & Gynecology at Ziekenhuis Oost-Limburg (ZOL) in collaboration with the Department of Physiology of Hasselt University in the framework of the Limburg Clinical Research Center (LCRC). CAPROM aims at evaluating the relationship between longitudinal (clinical) blood pressure measurements and changes in (subclinical) cardiovascular (CV) hemodynamics throughout pregnancy, as well as their responses to antihypertensive medication. To this end, CV profiling will be performed longitudinally on pregnant women at risk for developing GHD being included in the TM group of the PREMOM II study (group 1) or being followed-up via TM as part of their usual care (group 2). A separate ICF is signed for inclusion in the CAPROM substudy. The results of the CAPROM study will be performed by a researcher who is not involved in the PREMOM II main study. In addition, results of the CV profiling will not be communicated to the clinical decision makers of PREMOM II.

ELIGIBILITY:
Inclusion Criteria:

* a risk > 1/100 on the Fetal Medicine Foundation (FMF) tool, which is used from the following website: https://fetalmedicine.org/research/assess/preeclampsia/first-trimester
* CAPROM substudy: Pregnant women at risk for the development of GHD being followed-up via TM as part of the PREMOM II study (group 1) or usual care (group 2)

Exclusion Criteria:

* congenital malformations of the newborn,
* pregnant women who doesn't have a Smartphone,
* pregnant women < 18 years old,
* pregnant women who doesn't understand the Dutch/French/English language. -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Gestational age (GA) | Throug study completion, from the first contact with the gynaecologist (after fertilization) untill 34 weeks of gestation.
  difference of at least 10 days between the TM group and the CC was observed in our pilot studies, and will be used as a clinically relevant difference. An extension of the GA by even one day has a large impact on clinical outcomes for the neonate (both short- as long term). Moreover, the highest cost reductions were obtained in the group that delivered before 34 weeks of GA.
hospitalization | From 32 weeks of gestation until 34 weeks of gestation
  Numbers of hospitalization during pregnancy (Numeric. Available by hospital details of every patient who is included in the study. From the moment of hospitalization until the moment of discharge is 1 hospitalization.
Changes in CV physiological parameters - electrocardiogram (ECT) with Doppler ultrasonography | Month 3 to month 9
  The CV profile assessment consists of a simple, non-invasive method using the ECG with Doppler ultrasonography providing information about arteries and veins
changes in CV physiological parameters - impedance cardiography | Month 3 to month 9
  The CV profile assessment consists of a simple, non-invasive method using Impedance Cardiography using the Non-Invasive Continuous Cardiac Output (NICCOMO) monitor registering heart parameters
changes in CV physiological parameters - bio impedance | Month 3 to month 9
  The CV profile assessment consists of a simple, non-invasive method using Bio-Impedance using the Maltron® Bioscan 920-II giving information about the fluid balance.
Arterial parameters - pulse transit time | Month 3 to month 9
  The Pulse Transit Method (PTT) as a non-invasive means to track Blood Pressure over a short period of time
Arterial parameters - pulsatility index | Month 3 to month 9
  Pulsatility index (PI) is defined as the difference between the peak systolic flow and minimum diastolic flow velocity, divided by the mean velocity recorded throughout the cardiac cycle. It is a non-invasive method of assessing vascular resistance with the use of Doppler ultrasonography.
Arterial parameters - resistivity index of the left and right arcuate arteries | Month 3 to month 9
  The arterial resistive index is a sonographic index of intrarenal arteries defined as (peak systolic velocity - end-diastolic velocity) / peak systolic velocity. The normal range is 0.50-0.70.
venous parameters - venous pulse transit time of the hepatic and left and right renal veins | Month 3 to month 9
  Maternal venous pulse transit times (VPTT) weredefined as the time interval (ms) between the maternalECG P-wave and corresponding Doppler A-wave, correctedfor the duration of the corresponding cardiac cycle
venous parameters - hepatic vein impedance index | Month 3 to month 9
  ECG-Doppler parameters were impedance index at the level of hepatic veins (HVI) and renal interlobar veins (RIVI) together with venous pulse transit times (VPTT), as well as resistive and pulsatility index, and arterial pulse transit time (APTT) at the level of uterine arcuate arteries.
venous parameters - left and right renal interlobar vein impedance indices | Month 3 to month 9
  ECG-Doppler parameters were impedance index at the level of hepatic veins (HVI) and renal interlobar veins (RIVI) together with venous pulse transit times (VPTT), as well as resistive and pulsatility index, and arterial pulse transit time (APTT) at the level of uterine arcuate arteries.
systolic blood pressure | Month 3 to month 9
  systolic blood pressure (mmHg),
diastolic blood pressure | Month 3 to month 9
  diastolic blood pressure (mmHg),
Mean arterial blood pressure | Month 3 to month 9
  Mean arterial blood pressure (mmHg),
Total body water | Month 3 to month 9
  Total body water (liters)
extracellular water | Month 3 to month 9
  extracellular water (liters)
intracellular water | Month 3 to month 9
  intracellular water (liters)
ECW/ICW ratio | Month 3 to month 9
  ECW/ICW ratio
stroke volume | Month 3 to month 9
  stroke volume (ml)
hear rate (beats/min) | Month 3 to month 9
  hear rate (beats/min)
cardiac output (l/min) | Month 3 to month 9
  cardiac output (l/min)
velocity index (1/1,000/s) | Month 3 to month 9
  velocity index (1/1,000/s)
acceleration index (1/100/s²) | Month 3 to month 9
  acceleration index (1/100/s²)
total peripheral resistance (dyn·s·cm-5) | Month 3 to month 9
  total peripheral resistance (dyn·s·cm-5)

SECONDARY OUTCOMES:
number of prenatal consults | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  prenatal follow- up, numeric value, every consult during pregnancy from the first consultation until delivery
number of ultrasounds | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric value, every ultrasound during pregnancy from the first consultation until delivery
number of CTG's | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric value, every CTG during pregnancy from the first consultation until delivery
number of hospitalizations of the mother at the MIC department | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric value, every hospitalization at the MIC during pregnancy from the first consultation until delivery
number of days admitted to the MIC | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric value, amount of days admitted to the MIC from the first consultation unitil delivery
number of medication adaptations during pregnancy | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric value, every change from no medication intake/a specific medciation at a specific dose to another medication intake at a specific dose.
development of gestational hypertensive disorders | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric, the diagnoses of gestational hypertension/pre-eclampsia/HELLP during pregnancy
Onset of delivery | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  categorical (spontaneous, induced, primary section) from birth until discharge from the hospital
Mode of delivery | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  categorical (vaginal, instrumental, primary/secondary section) from birth until discharge from the hospital
Birthweight | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  gram from birth until discharge from the hospital
Apgar at 1' and 5' | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric (0-10) from birth until discharge from the hospital
Admission to the neonatal intensive care (NIC) | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  categorical(Yes/no) from birth until discharge from the hospital
Number of days admitted to the NIC | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric value, amount of days admidtted to the NIC, from birth until discharge from the hospital
Cost for the health care services (HCS) | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  Costs of the prenatal care as described in Secondary outcomes (1) and costs for the care during and after the delivery as described in Secondary outcomes (2), which are divided in: costs for the HCS, costs for the patient, costs for the RIZIV. All costs will be collected in Euros. rom the first contact with the gynaecologist until the discharge from the hospital of both the mother and the neonate.
number of phone calls from the patient to the midwife for technical issues | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric scale, contributor to the added value of TM
number of phone calls from the patient to the midwife for medical issues | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric scale, contributor to the added value of TM
number of phone calls from the midwife to the patient for technical issues | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric scale, contributor to the added value of TM from the inclusion in the study until the moment of delivery
number of phone calls from the midwife to the patient for medical issues | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric scale, contributor to the added value of TM from the inclusion in the study until the moment of delivery
number of starts/adjustments to the antihypertensive medication | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  numeric scale, contributor to the added value of TM from the inclusion in the study until the moment of delivery
Changes in CV profile throughout pregnancy and in response to medication | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  Changes in Cardiovascular profile throughout pregnancy and in response to medication
BMQ questionaire | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  Beliefs about Medicine Questionnaire
ProMAS Questionnaire | during pregnancy from the first consultation until delivery assessed up to 40 weeks
  a Probabilistic Medication Adherence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Gyselaers, prof. dr., Principal Investigator — Hasselt University; Dorien Lanssens, dr., Study Chair — Hasselt University
Locations (5):
- Belgium (5):
  - University hospital Antwerp, Antwerp
  - AZ Sint-Lucas Brugge - Oostende, Bruges
  - AZ Sint Jan Brugge - Oostende, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - Universitaire Ziekenhuizen Leuven, Leuven

REFERENCES:
- [Derived] Dreesen P, Lanssens D, Nouwen S, Volders P, Janssen F, Soubry A, Gyselaers W, Ceulemans M. Medication beliefs and adherence during and after pregnancy among women at risk for gestational hypertensive disorders. Front Drug Saf Regul. 2025 Aug 11;5:1610273. doi: 10.3389/fdsfr.2025.1610273. eCollection 2025. PMID 40978500
- [Derived] Lanssens D, Thijs IM, Gyselaers W; PREMOM II - consortium. Design of the Pregnancy REmote MOnitoring II study (PREMOM II): a multicenter, randomized controlled trial of remote monitoring for gestational hypertensive disorders. BMC Pregnancy Childbirth. 2020 Oct 15;20(1):626. doi: 10.1186/s12884-020-03291-2. PMID 33059633
- [Derived] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394